CLINICAL TRIAL: NCT00728130
Title: Prospective Study to Assess the Anatomical Relationship of Level IB Lymph Nodes to the Submandibular Gland in Patients With Carcinoma of the Upper Aerodigestive Tract
Brief Title: Anatomical Relationship of Level IB Lymph Nodes to the Submandibular Gland in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RON-SCCI 08-003-1
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Results first posted 2013-07-29 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Carcinoma
Keywords: carcinoma; upper; aerodigestive; tract; submandibular; gland
MeSH Terms: conditions — Carcinoma | interventions — iso-sulfan blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): A neck dissection of at least the ipsilateral sub-level 1B will be performed in all patients
  Interventions: Procedure: neck dissection of at least the ipsilateral sub-level 1B

INTERVENTIONS:
Procedure: neck dissection of at least the ipsilateral sub-level 1B — neck dissection of at least the ipsilateral sub-level 1B
  Other Names: Lymphazurin®

SUMMARY:
Hypothesis

1. The submandibular gland is not a lymphatic organ and usually remains uninvolved with head and neck cancer despite the presence of metastatic disease in the lymph nodes that surround it.
2. All the lymph nodes in the submandibular triangle can be removed without resection of the submandibular gland.

Study Design

A better understanding of the frequency of submandibular gland involvement may lead to refined treatment strategies for head and neck cancer, which can possibly spare removal of the submandibular gland and potentially improve the long term side effects from therapy.

DETAILED DESCRIPTION:
Hypothesis

1. The submandibular gland is not a lymphatic organ and usually remains uninvolved with head and neck cancer despite the presence of metastatic disease in the lymph nodes that surround it.
2. All the lymph nodes in the submandibular triangle can be removed without resection of the submandibular gland.

Study Design

1. A prospective controlled study.
2. A neck dissection of at least the ipsilateral sub-level 1B will be performed in all patients. In case of oral cavity tumors, about 15 minutes prior to the surgery, 1ml of Lymphazurin® blue dye will be injected in 4 quadrants around the primary site. The dissection will be performed in 3 stages. In the first stage all lymph node groups that lie either lateral, anterior, posterior, superior, or inferior to the submandibular gland, but within anatomical boundaries of level 1B, will be dissected. The submandibular gland will be left intact for this portion of the procedure. Next, the submandibular gland will be removed. Lastly, any remaining fibrofatty tissue that lies deep to the submandibular gland within the confines of level IB will be removed. Each lymph node group, the submandibular gland, and the fibrofatty tissue lying deep to the submandibular gland, will be submitted for pathological assessment in separate containers.
3. The following end-points will be measured: the number of lymph nodes identified within each lymph node group, the number of lymph nodes located within the submandibular gland, and the number of lymph nodes within the fibrofatty contents lying deep to the submandibular gland. The presence or absence of carcinoma within each of the assessed nodes will be documented, as well as extracapsular spread.

A better understanding of the frequency of submandibular gland involvement may lead to refined treatment strategies for head and neck cancer, which can possibly spare removal of the submandibular gland and potentially improve the long term side effects from therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed carcinoma of the oral cavity, oropharynx, larynx or hypopharynx
* Treatment of the regional lymph nodes to include neck dissection performed as the primary modality
* No previous treatment to the neck
* No previous treatment for the index cancer (surgery, chemotherapy, radiation or biological therapy)
* No known distant metastatic disease
* Age >/= 18
* The ability to understand and willingness to sign a study-specific written informed consent form
* Protocol treatment must begin </= 8 weeks of diagnostic biopsy

Exclusion Criteria:

* Previous or concurrent head and neck primaries
* Prior surgery to study site other than biopsy
* Patients receiving any other treatment for cancer within 30 days previously
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements
* Known allergy to Lymphazurin®
* Pregnant or breast feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Robbins, M.D., Principal Investigator — SIU School of Medicine
Locations (1):
- SIU School of Medicine, Springfield, Illinois, United States

REFERENCES:
- [Background] Robbins KT, Clayman G, Levine PA, Medina J, Sessions R, Shaha A, Som P, Wolf GT; American Head and Neck Society; American Academy of Otolaryngology--Head and Neck Surgery. Neck dissection classification update: revisions proposed by the American Head and Neck Society and the American Academy of Otolaryngology-Head and Neck Surgery. Arch Otolaryngol Head Neck Surg. 2002 Jul;128(7):751-8. doi: 10.1001/archotol.128.7.751. No abstract available. PMID 12117328
- See also: sponsoring institution website — http://www.siumed.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment planning was performed for all patients in the multidisciplinary head and neck oncology forum before recruitment into the trial.
  Dates of recruitment: 06/11/2008 through 09/17/2009 Number of patients recruited: 23 Number of patient completing trial: 20
Groups:
- Surgery: A neck dissection of at least the ipsilateral sub-level 1B will be performed in all patients.
Period: Overall Study
Arm/Group | Surgery
Started | 22
Completed | 19
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Paperwork not completed in time | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Surgery
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (10.8)
Age, Customized [Number; unit: participants]
  <=18 years | 0
  Between 18 and 79 years | 22
  >=80 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14
submandibular gland excision [Number; unit: participants]
  Surgery | 19
  Not completed | 3
sublevel IB dissection [Number; unit: participants]
  Surgery | 19
  Not completed | 3
surgical bed inspection [Number; unit: participants]
  Surgery | 19
  Not completed | 3

OUTCOME MEASURES:

1. Primary Outcome: the Number of Lymph Nodes: 1. Identified Within Each Lymph Node Group, 2.Located Within the Submandibular Gland, and 3. Within the Fibrofatty Contents Lying Deep to the Submandibular Gland.
Description: The number of head/ neck lymph nodes in pre-defined groups: Preglandular, Prevascular, Retrovascular, and Retroglandular as well as the number of nodes within the submandibular gland and within the fibrofatty contents lying deep to the submandibular gland.
Time Frame: Post Surgical Time point
Measure: Mean (Standard Deviation); unit: nodes
Groups:
- Surgical Lymph Node Groups: A neck dissection of at least the ipsilateral sub-level 1B will be performed in all patients. The number of nodes for each nodal groups will be reported.
Arm/Group | Surgical Lymph Node Groups
Number analyzed (Participants) | 19
nodes
  Preglandular nodal group-Right neck | 2.3 (1.4)
  Prevascular nodal group-Right neck | 1.1 (0.8)
  Retrovascular nodal group-Right neck | 1.0 (1.3)
  Retroglandular nodal group-Right neck | 1.1 (1.1)
  Preglandular nodal group-Left neck | 1.5 (1.3)
  Prevascular nodal group-Left neck | 2.3 (1.7)
  Retrovascular nodal group-Left neck | 1.4 (1.5)
  Retroglandular nodal group-Left neck | 1.1 (1.2)
  Submandibular nodes (Right or Left) | 0 (0)
  Nodes Deep to Submandibular gland (Right or Left) | 0 (0)

2. Secondary Outcome: The Presence or Absence of Carcinoma Within Each of the Assessed Nodes Will be Documented, as Well as Extracapsular Spread.
Description: Pathological detection of carcinoma within each of the dissected nodes reported as node groups.
Time Frame: Post surgical time point
Measure: Mean (Standard Deviation); unit: carcinoma positive nodes
Arm/Group | Surgical Lymph Node Groups
Number analyzed (Participants) | 19
carcinoma positive nodes
  Preglandular nodal positivity right neck | 0 (0)
  Prevascular nodal positivity right neck | 0.1 (0.8)
  Retrovascular nodal positivity right neck | 0 (0)
  Retroglandular nodal positivity right neck | 0 (0)
  Preglandular nodal positivity left neck | 0.2 (0.6)
  Prevascular nodal positivity left neck | 0.3 (0.6)
  Retrovascular nodal positivity left neck | 0 (0)
  Retroglandular nodal positivity left neck | 0 (0)

ADVERSE EVENTS:
Arm/Group | Surgery
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No